CLINICAL TRIAL: NCT06161103
Title: Comparison of the Clinical Success of 3D Printed Prefabricated Composite Resin Crowns With Stainless Steel Crowns: A Randomised Controlled Trial
Brief Title: Comparison of 3D Printed Composite Resin Crowns With Stainless Steel Crowns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUPediatricDentistry 3D Crown
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Carious Teeth
Keywords: 3D printing, stainless steel crowns, composite resin crowns
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 3D Printed Prefabricated Composite Resin Crown group (Experimental): (Custom Composite Resin (Custom Resin Solutions, CRSCAM TEKNOLOJİ AŞ., ANTALYA, TURKEY)
  Interventions: Procedure: 3D Printed Prefabricated Composite Resin Crown Group
- Active Comparator: Prefabricated stainless steel crown group (Experimental): Stainless Steel Crown (SSC, Kids Crown, Shinghung, Seoul, Korea)
  Interventions: Procedure: Prefabricated stainless steel crown group

INTERVENTIONS:
Procedure: 3D Printed Prefabricated Composite Resin Crown Group — 3D Crown application: After preparing the molars, the crown was cemented by passive seating with modified glass ionomer cement (GC FujiCEM Evolve, GC America, Alsip, USA).
  Arms: Experimental: 3D Printed Prefabricated Composite Resin Crown group
Procedure: Prefabricated stainless steel crown group — Stainless steel crown application: After preparing the molars, the crown was filled with type-1 glass ionomer cement (Aqua Meron, Voco, Cuxhaven, Germany) and cemented.
  Arms: Active Comparator: Prefabricated stainless steel crown group

SUMMARY:
The goal of this splith - mouth clinical trial is to compare 3D Printed Prefabric Composite Resin Crowns with Stainless Steel Crowns in healthy 50 children age between 5 and 9 with caries on more than one surface of the primary second molars.

The main question[s] it aims to answer are:

* 3D printed composite resin crown's survival rate is as succesful as stainless steel crowns
* 3D printed composite resin crowns periodontal integrity is as succesful as stainless steel crowns

Condition or disease : Carious Teeth

Intervention/treatment:

Procedure/Surgery: 3D Printed Prefabricated composite resin crown group Procedure/Surgery: Prefabricated stainless steel crown group

DETAILED DESCRIPTION:
In this study, 3D Printed prefabricated composite resin crowns will be compared with prefabricated stainless steel crowns in a randomized controlled manner. The study will be conducted in split-mouth to eliminate the effect of potential confounders. The obtained data will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 5-9 years with caries on second primary molars
* Children without systemic disease or developmental dental anomalies that may affect caries susceptibility.
* Children whose cooperation is 'positive' or 'absolutely positive' according to the Frankl behavioral scale (Frankl et al., 1962).
* Those with deep dentin caries that do not extend to the pulp in the teeth to be treated
* The molars will be treated with a crown indication.
* Presence of symmetry of the primary molar to be treated in the opposite arch.
* The molar to be treated is in occlusion with the antagonist.
* Presence of caries on at least two surfaces of the molars to be treated.
* Absence of spontaneous pain, abscess, mobility, interradicular lesion in the tooth to be treated
* Patients whose parents and themselves agree to participate in the treatment

Exclusion Criteria:

* Children whose treatment cannot be continued on the dental chair due to cooperation
* Molars that will soon be exfoliated, 1/2 of the root has been resorbed
* The presence of bruxism
* The presence of erosion or attrition-related wear on the opposing molar
* The patient does not come to the control appointment or does not want to continue to the research
* Have allergy to local anesthetic, nickel or chromium
* Complications during treatment.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinical success | 24 Month
  According to the criteria reported by Santamaria et al. (2004), clinical success will be categorized as successful, major failure, and minor failure.
  Successful:
  No clinical signs or symptoms of pulp pathology Tooth has exfoliated (without any minor/major failures) No deformations in the crown/restoration No pathology observed in radiographs
  Minor failure:
  Reversible pulpitis (No need for root canal treatment or extraction) Crown/restoration loss that can be restored Presence of deformations/fractures/perforations in the crown/restoration Permanent crown remaining submerged Presence of new caries at the margins
  Major failure:
  Irreversible pulpitis Crown/restoration loss that cannot be restored Inter-radicular radiolucency Internal root resorption
United States Public Health Service (USPHS): Retention, marginal compliance and gingival health criteria | 24 Month
  Restorations were evaluated to determine success according to modified United States Public Health Service (USPHS) criteria for marginal adaptation, marginal discolouration, secondary caries, anatomical form, retention, postoperative sensitivity and colour matching. Restorations with an "Alpha (A)" score were considered successful, those with a "Bravo (B)" score were considered acceptable, and those with a "Charlie (C)" score were considered unsuccessful. The scoring of the restorations was decided by agreement of both dentists (Ryge G. et al., 1980).
Marginal Crown Gap | 24 Month
  (0) ¼ at the gingival margin, (1) ¼ below the gingival line (apical to the gingival margin) or (2) ¼ above the gingival line (occlusal to the gingival margin) [Muhamed Altinawia et al., 1980].
Plaque Index (PI) (Silness and Loe, 1964) | 24 Month
  In this index, the thickness of dental plaque on the mesial, distal, vestibular, lingual tooth surfaces of all teeth or selected teeth and in relation to the gingiva is evaluated by probing. The values determined on the surfaces are summed and the plaque index value of the individual is obtained by taking the mathematical average.
  0-No plaque in the area adjacent to the gingiva
  1. There is a thin film on the edge of the gingival margin. This formation can only be detected with the help of a probe.
  2. There is plaque in the gingival pocket and gingival margin at a level that can be determined by eye. There is no plaque in the aproximal area.
  3. A large amount of plaque layer is observed in the gingival pocket and gingival margin. Interdental areas are filled with plaque.
Gingival Index (GI) (Löe & Silness, 1963) | 24 Month
  It evaluates bleeding, which is the most basic sign of inflammation. The mesial, distal, vestibule and lingual sides of the teeth are evaluated. These values are then summed and divided by four.
  0- Healthy gingiva, no inflammation
  1. Mild inflammation, discolouration and mild oedema of the gums, no bleeding on probing
  2. Moderate inflammation, redness and oedema of the gums, bleeding on probing
  3. There is advanced inflammation, redness, oedema in the gum, spontaneous bleeding is observed.
Simplified Oral Hygiene Index (OHI-S) | 24 Month
  Simplified Oral Hygiene Index (OHI-S) will be used to evaluate the plaque and calculus deposits of the patient and control groups. In this index, in order to simplify the oral hygiene index, six index teeth, which are considered representative of all anterior and posterior teeth, are evaluated. These teeth are teeth numbered 16, 26, 11, 31, 36, 46. The facial surfaces of teeth 16-26-11-31 and the lingual surfaces of teeth 36-46 are evaluated. This facilitation process is used both in the calculation of the debris index and in the calculation of the calculus index. After calculating the debris and calculus assessment indices, a simplified oral hygiene index is obtained (REF: 29.Greene, J.C., Vermillion, J.R.: The Simplified Oral Hygiene Index, J. Amer. Dent. Ass 68 : 7, 1960).
  The Simplified Oral Hygiene Index (OHI-S) Debris Index 0- No debris.
  1. There is debris less than 1/3 of the tooth surface.
  2. There is debris more than 1/3 and less than 2/3 of the tooth surface.
  3. More

IPD SHARING:
Plan to Share IPD: No